CLINICAL TRIAL: NCT02860052
Title: A Phase 2 Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Dose-Ranging Study Assessing Efficacy and Safety of SB208 and Vehicle Gel in Subjects With Interdigital Tinea Pedis
Brief Title: SB208 for the Treatment of Tinea Pedis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AF201
Record Dates: First submitted 2016-08-02; First posted 2016-08-09 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-11

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SB208 2% (Experimental): Apply once daily to one or both feet for 14 days
  Interventions: Drug: SB208 2%
- SB208 4% (Experimental): Apply once daily to one or both feet for 14 days
  Interventions: Drug: SB208 4%
- SB208 16% (Experimental): Apply once daily to one or both feet for 14 days
  Interventions: Drug: SB208 16%
- Vehicle Gel (Placebo Comparator): Apply once daily to one or both feet for 14 days
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: SB208 2% — Apply once daily to one or both feet for 14 days
  Other Names: NVN1000 4%
  Arms: SB208 2%
Drug: SB208 4% — Apply once daily to one or both feet for 14 days
  Other Names: NVN1000 8%
  Arms: SB208 4%
Drug: SB208 16% — Apply once daily to one or both feet for 14 days
  Other Names: NVN1000 32%
  Arms: SB208 16%
Drug: Vehicle Gel — Apply once daily to one or both feet for 14 days
  Other Names: Vehicle
  Arms: Vehicle Gel

SUMMARY:
This is a phase 2, multi-center, double-blind, randomized, vehicle-controlled study to be conducted in non immunocompromised adult subjects with interdigital tinea pedis.

DETAILED DESCRIPTION:
A phase 2, multi-center, double-blind, randomized, vehicle-controlled study to be conducted in approximately 170 non immunocompromised adult subjects with interdigital tinea pedis. Subjects will apply the investigational product (IP) (SB208 or Vehicle Gel) to the interdigital areas and all affected and immediate surrounding areas of one or both feet once daily for 2 weeks, followed by a 4-week post-treatment observation period.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male and female subjects with clinical diagnosis of interdigital t. pedis
* T.pedis provisionally confirmed at baseline by a positive KOH wet mount for segmented fungal hyphae on skin scraping from the target site

Exclusion Criteria:

* Women who are pregnant or nursing or planning on becoming pregnant
* Subjects with onychomycosis or moccasin-type t. pedis
* Subjects using topical or systemic anti-fungal agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Fungal culture result | 2 weeks
  Negative fungal culture from target lesion

SECONDARY OUTCOMES:
Clinical cure | 6 wks
  Amelioration of signs and symptoms of tinea pedis
Mycological cure | 6 wks
  No evidence of fungal infection based on skin scraping and culture

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events | 6 weeks
  Summary of treatment emergent adverse events by treatment group

CONTACTS AND LOCATIONS:
Overall Officials: M Joyce Rico, MD, Study Director — Novan, Inc.
Locations (1):
- Instituto Dermatológico y Cirugía de Piel,, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No